CLINICAL TRIAL: NCT02720406
Title: Topical Ketamine by Neubulization Method in Tonsillectomy
Brief Title: Topical Ketamine Analgesia in Children Undergoing Tonsillectomy: a Clinical and Serum Level Assays Study.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AssuitUniversity
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intravenous ketamine0.5mg/kg (Active Comparator): intravenous ketamine 0.5 mg/kg given after induction of anesthesia and before surgery.
  Interventions: Drug: Intravenous ketamine0.5mg/kg
- Nebulized ketamine 1mg/kg (Active Comparator): nebulized ketamine group received 1mg/kg ketamine by nebulzation before induction of anesthesia.
  Interventions: Drug: Nebulized Ketamine 1mg/kg
- Nebulized ketamine 2mg/kg (Active Comparator): nebulized ketamine group received 2mg/kg ketamine by nebulzation before induction of anesthesia.
  Interventions: Drug: Nebulized Ketamine 2mg/kg
- control group (Placebo Comparator): control group received placebo nebulization
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: Intravenous ketamine0.5mg/kg — Intravenous ketamine 0.5mg/kg after anesthesia and before surgery.
  Other Names: Katalar
  Arms: Intravenous ketamine0.5mg/kg
Drug: Nebulized Ketamine 1mg/kg — Nebulized Ketamine 1mg/kg given by nebulizer before anesthesia.
  Other Names: Katalar
  Arms: Nebulized ketamine 1mg/kg
Drug: Nebulized Ketamine 2mg/kg — Nebulized Ketamine 2mg/kg given by nebulizer before anesthesia.
  Other Names: Katalar
  Arms: Nebulized ketamine 2mg/kg
Drug: saline placebo — Saline 0.9% given by nebulizer before anesthesia and iv after anesthesia and before surgery.
  Other Names: Saline
  Arms: control group

SUMMARY:
The aim of this study is to evaluate the analgesia efficacy of local ketamine given by two different doses in pediatric patients undergoing tonsillectomy operations

DETAILED DESCRIPTION:
In this double-blinded, clinically-controlled trial, 100 child will be randomized into four groups of 25 patients each; control group, intravenous ketamine group received 0.5mg iv. ketamine, and two local ketamine groups receiving local ketamine by nebulization in two different doses; 1 and 2mg/kg. The verbal rating pain scale, time to first postoperative analgesic request, total analgesic consumption during 1st 24 h postoperative, serum ketamine levels, intra operative blood loss, postoperative bleeding, and adverse effects were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients aged 7-12 years and scheduled for elective tonsillectomy due to recurrent or chronic tonsillitis will be included in the study

Exclusion Criteria:

* patients with known hypersensitivity to medication drugs, coagulation disorders, thrombocytopenia, and significant cardiac, renal, pulmonary or hepatic disease.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | 24 hours postoperative
  The total amount of analgesics used in the first 24h postoperative in mg.

SECONDARY OUTCOMES:
Postoperative pain scores | 24 hours postoperative
  Pain intensity will be assessed postoperatively by using the Verbal Rating scale (VRS) (0 =no pain, 1 =mild pain, 2 =moderate pain, 3 =severe pain, and lastly 4 =excruciating pain). VRS assessments were performed at rest in the following time points; at arrival to PACU, 30 min, 1, 2, 3, 4, 5, 6, 12, and 24 h postoperative.
  -
  -
  .
Ketamine serum levels to exclude systemic absorption of topical ketamine. | 120 min after receiving Ketamine
  the level of ketamine in the serum.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No